CLINICAL TRIAL: NCT01328457
Title: An Effectiveness Study of Paromomycin IM Injection (PMIM) for the Treatment of Visceral Leishmaniasis (VL) in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Shaheed Suhrawardy Medical College Hospital, Dhaka, Bangladesh (Unknown); GVK Biosciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VLPMIM402
Record Dates: First submitted 2011-01-21; First posted 2011-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2012-08

CONDITIONS: Visceral Leishmaniasis
Keywords: Leishmaniasis, Visceral; kala-azar; Paromomycin; Bangladesh; Injections, Intramuscular; Treatment Outcome; Patient compliance; Medication adherence; Drug toxicity
MeSH Terms: conditions — Leishmaniasis, Visceral; Patient Compliance; Medication Adherence; Drug-Related Side Effects and Adverse Reactions | interventions — Paromomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Paromomycin sulfate — Paromomycin IM Injection, 11 mg/kg as the base, intramuscular, once a day on 21 consecutive days (or no more than 22 days if one injection is missed during the treatment period).
  Other Names: aminosidin sulfate; aminosidine sulfate; monomycin A sulfate; amminosidin sulfate; catenulin sulfate; crestomycin sulfate; estomycin sulfate; hydroxymycin sulfate; neomycin E sulfate; paucimycin sulfate; Humatin®; Gabbromicina®; Gabromicina®; Gabromycin®; Gabboral®; Kapseal®; Pargonyl

SUMMARY:
The purpose of this study is to evaluate the effectiveness of treatment with PMIM in patients with visceral leishmaniasis within the VL-endemic region of Bangladesh at EOT (21/22 days after treatment begins), and at 6 months after end of treatment (Day 202/203, -15 to +30 days).

DETAILED DESCRIPTION:
Safe, effective and affordable treatments for visceral leishmaniasis (VL) that are widely available to the poorest populations are urgently needed in Bangladesh in areas where the disease is endemic. Paromomycin IM Injection (PMIM) was approved for the treatment of VL in August 2006 by the Drugs Controller General of India (DCGI), and it offers an attractive alternative to treatments that are currently available.

ELIGIBILITY:
Inclusion Criteria:

1. Signs and symptoms of VL including:

   * History of intermittent fever for at least two weeks
   * History of weight loss and/or decrease in appetite
   * Enlarged spleen
2. VL serologically confirmed using the rK39 test:
3. Willingness / ability to understand and provide informed consent prior to participation in this study:
4. Age ≥ five years and ≤ 55 years, and weighing at least five kg
5. Adequately hydrated as assessed by clinical criteria and able to maintain adequate hydration on an outpatient basis through oral intake of fluids
6. Clinically stable and appropriate for treatment with PMIM as an outpatient, if possible (subjects may be hospitalized to receive 21-day dosing at the discretion of the investigator)
7. Living in the VL-endemic areas in Bangladesh

Exclusion Criteria:

1. Active tuberculosis or taking anti-tuberculosis medications
2. Previous treatment with Paromomycin IM Injection (PMIM)
3. Clinically significant severe anemia as determined by the investigator
4. Clinically significant renal or hepatic dysfunction as determined by the investigator, or history of clinically significant renal or hepatic dysfunction
5. History of Hepatitis B or C; or known HIV positive
6. History of hearing loss
7. Other serious illness or medical condition that, in the opinion of the doctor, would interfere with the patient's ability to receive PMIM treatment or comply with the study procedures, or that could obscure toxicity of or response to PMIM
8. Major surgery within 30 days prior to first dose of PMIM
9. History of hypersensitivity to aminoglycosides or to any of the components of PMIM, including sulfite
10. Any history of VL or treatment of VL at any time
11. Patients who have received any investigational (unlicensed) drug within the last six months
12. Concomitant use of other aminoglycosides (e.g., gentamicin, tobramycin, amikacin), nephrotoxic and ototoxic drugs, or immunosuppressive drugs
13. Proteinuria (results > 1+ ) on urine dipstick analysis at screening visit and/or
14. Serum creatinine above the upper limit of normal (ie, serum creatinine >1.1 mg/dl in males and >0.9 mg/dl in females
15. Pregnant or lactating women

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Final cure rate | 6 months after end of treatment (Day 202/203, -15 to +30 days)
  Criteria evaluated (binary fashion):
  1. Patient's temperature less than 99.4°F in clinic at EOT visit? (Y/N)
  2. Patient reported resolution of fever and NO fever within the last 5 days? (Y/N)
  3. Spleen size decreased from screening value? (Y/N)
  4. Is the clinical impression of the treating physician that of an adequate clinical response? (Y/N)
  The patient is deemed to have achieved final cure if answers to a, b, c, AND d are all "Yes" OR if one answer (a, b, or c) is "No" but all others and "d" are "Yes". In addition, the clinician will inquire about pregnancy status for female patients.

SECONDARY OUTCOMES:
Initial clinical response rate | End of treatment (21/22 days after treatment begins)
  Criteria evaluated (binary fashion):
  1. Patient's temperature less than 99.4°F in clinic at EOT visit? (Y/N)
  2. Patient reported resolution of fever / NO fever within the last 5 days? (Y/N)
  3. Spleen size decreased from screening value? (Y/N)
  4. Is clinical impression of the treating physician that of an adequate clinical response? (Y/N)
  The patient is deemed to achieve an initial clinical response if answers to a, b, c, AND d are all "Yes" OR if one answer (a, b, or c) is "No" but all others and "d" are "Yes". Also, the clinician will inquire re: pregnancy status for female patients.
Patient compliance with PMIM treatment | 22 days
  Proportion of patients complying with prescribed 21 daily injections over no more than 22 days.
Safety of PMIM in the study population based on clinical assessment by the study physician at the Upazilla Health Centre. | 6 months after end of treatment
  All serious adverse events (SAEs), regardless of causality, from time of first administration of PMIM through 30 days post-EOT.
  All adverse events (AEs), regardless of causality, from time of first dose through 30 days post-EOT.
  Vital signs on Study Days 1 to 21/22 (or early termination), any unscheduled visit after EOT, 30 days after EOT, and 6 months after EOT.
  Patients who become pregnant during treatment/within 30d following EOT will be included in the safety population. Offspring from pregnancies will be followed for safety under a separate study for a period up to 3 yrs after birth.
To introduce PMIM in government health facilities in rural Bangladesh. | October 2011
  Training study staff to provide treatment with PMIM at selected Upazila level health complexes in rural Bangladesh.

CONTACTS AND LOCATIONS:
Overall Officials: Rashidul Haque, MB, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (3):
- Bangladesh (3):
  - Bhaluka Upazila Health Complex, Bhaluka, Mymensingh District
  - Trishal Upazila Health Complex, Trishal, Mymensingh District
  - Icddr,B, Dhaka

REFERENCES:
- [Background] Sundar S, Jha TK, Thakur CP, Sinha PK, Bhattacharya SK. Injectable paromomycin for Visceral leishmaniasis in India. N Engl J Med. 2007 Jun 21;356(25):2571-81. doi: 10.1056/NEJMoa066536. PMID 17582067
- [Background] Kanyok TP, Killian AD, Rodvold KA, Danziger LH. Pharmacokinetics of intramuscularly administered aminosidine in healthy subjects. Antimicrob Agents Chemother. 1997 May;41(5):982-6. doi: 10.1128/AAC.41.5.982. PMID 9145856
- [Derived] Jamil KM, Haque R, Rahman R, Faiz MA, Bhuiyan AT, Kumar A, Hassan SM, Kelly H, Dhalaria P, Kochhar S, Desjeux P, Bhuiyan MA, Khan MM, Ghosh RS. Effectiveness Study of Paromomycin IM Injection (PMIM) for the Treatment of Visceral Leishmaniasis (VL) in Bangladesh. PLoS Negl Trop Dis. 2015 Oct 23;9(10):e0004118. doi: 10.1371/journal.pntd.0004118. eCollection 2015. PMID 26496648